CLINICAL TRIAL: NCT07356258
Title: Iron Supplementation Frequency and Tolerability in Pregnancy
Brief Title: Oral Iron in Pregnant Women: How Often to Take It and Its Side Effects and Tolerability
Acronym: IRONFIT
Status: Not yet recruiting | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: BNZ 013424
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Iron Adverse Reaction; Anemia Complicating Pregnancy
Keywords: pregnancy; iron tolerability; oral iron supplementation; ron deficiency anemia; ferrous sulfate; alternate-day dosing; daily dosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. It's an observational study — No intervention. It's an observational study

SUMMARY:
The goal of this prospective observational study is to examine the frequency of gastrointestinal side effects associated with oral iron supplementation during pregnancy. The main question it aims to answer is:

Does intermittent oral iron supplementation result in fewer gastrointestinal side effects compared with daily supplementation in pregnant women? Pregnant women who are prescribed oral iron as part of their routine medical care will take ferrous sulfate on an alternate-day schedule for one week. If no significant gastrointestinal side effects are reported, they will then take ferrous sulfate daily for an additional week and will be followed for one month. Participants will be contacted by the study investigator to report gastrointestinal side effects, and routine blood tests will be used to assess changes in hemoglobin and iron stores.

DETAILED DESCRIPTION:
This prospective observational study will be conducted in pregnant women who are prescribed oral iron supplementation as part of their routine prenatal care. The study is designed to reflect standard clinical practice and does not introduce any investigational treatment or deviation from accepted management.

Following enrollment, participants will receive oral ferrous sulfate in accordance with common clinical recommendations. The study includes two sequential exposure periods: an initial alternate-day dosing phase followed by a daily dosing phase, provided that no significant gastrointestinal intolerance is reported during the first phase.

At baseline, relevant demographic and pregnancy-related information will be recorded, including maternal age and gestational age at initiation of iron therapy. Baseline laboratory values related to iron status (including hemoglobin and iron stores) will be documented if obtained as part of routine care.

Participants will be instructed to take oral iron according to the prescribed schedule and to continue their usual diet and prenatal care. No dietary restrictions will be imposed as part of the study. Information regarding timing of iron intake, concomitant food consumption (including dairy products), and adherence will be collected through participant self-report.

Participants will be contacted by the study investigator at predefined time points during the supplementation period. Structured interviews will be used to assess gastrointestinal side effects, including constipation, abdominal pain, nausea, vomiting, diarrhea, bloating, and heartburn. Participants will be asked whether symptoms are new, worsened, or unchanged compared with baseline.

At one month after initiation of iron supplementation, participants will undergo follow-up blood tests as part of routine clinical monitoring to assess hemoglobin concentration and iron stores.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-50
* Indication for oral iron treatment as determined by the treating physician, in accordance with standard clinical practice
* Baseline iron store levels measured prior to initiation of oral iron therapy

Exclusion Criteria:

* Women taking ferrous sulfate 80 mg Tardiferon
* Gastrointestinal diseases such as colitis
* Women who received intravenous iron during pregnancy
* Women who received blood transfusions during pregnancy
* Women with anemia due to causes other than iron deficiency
* History of bariatric surgery
* Allergy to ferrous sulfate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women attending our high-risk pregnancy clinics (in Bnai Zion medical center)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of gastrointestinal side effects in response to iron intake | Over the first 2 weeks of supplementation, with structured follow-up at week 1 and week 2

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No